CLINICAL TRIAL: NCT00498069
Title: Feasibility Study of the Safety and Activity of Autologous Bone Marrow Aspirate Concentrate (BMAC) for the Treatment of Critical Limb Ischemia Due to Peripheral Arterial Occlusive Disease
Brief Title: Study of Autologous Bone Marrow Concentrate for the Treatment of Critical Limb Ischemia (CLI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvest Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2007-1
Record Dates: First submitted 2007-07-05; First posted 2007-07-09 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2014-06

CONDITIONS: Ischemia
Keywords: Critical limb ischemia due to peripheral arterial occlusive disease; Autologous bone marrow concentrate
MeSH Terms: conditions — Ischemia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Injection of autologous bone marrow concentrate into ischemic tissues of the lower extremity
  Interventions: Device: Harvest Smartprep2 BMAC System; Device: SmartPReP2 BMAC System
- 2 (Placebo Comparator): Injection of placebo into ischemic tissues of the lower extremity
  Interventions: Biological: placebo

INTERVENTIONS:
Device: Harvest Smartprep2 BMAC System — injection of 40cc bmac
  Other Names: SmartPReP2 BMAC System
  Arms: 1
Device: SmartPReP2 BMAC System — Injection of autologous bone marrow concentrate prepared with the SmartPReP2 BMAC System
  Arms: 1
Biological: placebo — injection of placebo into ischemic tissue of the lower extremity
  Arms: 2

SUMMARY:
Injections of concentrated bone marrow mononuclear cells into ischemic tissues will result in vasculogenesis

DETAILED DESCRIPTION:
Bone marrow aspirate is collected and processed by centrifugation to remove red blood cells. The buffy coat is concentrated by removing plasma. The resultant concentrate of cells is injected into ischemic tissues of the lower limb.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Critical Limb Ischemia per protocol (see diagnostic criteria #2) with regard to the study limb.

Existence of a PAOD with clinical presentation corresponding to Rutherford Category 4 or Category 5 as defined in the reporting standards adopted by the Society of Vascular Surgeons (table 1)

* Patient meets at least one of the following diagnostic criteria in the study limb:

  * Ankle artery occlusion pressure absolute <50 mmHg or ABI <0.4
  * Toe artery occlusive pressure < 40mm Hg or TBI (<0.4)
  * TcPO2 <20 mmHg lying down breathing room air.
* There is no reasonable open surgical or endovascular revascularization option as determined by the treating vascular specialist. Factors that may contribute to the determination of inoperability may include:

  * Anatomical considerations

    * No outflow targets
    * No appropriate conduit (i.e. vein for bypass)
    * Long segment occlusions or calcified lesions that predict poor outcome with endovascular approaches.
  * High risk medical conditions

    * Unstable cardiac disease.
    * Renal insufficiency
  * History of prior failed revascularization attempts
  * The patient's unsuitability must be confirmed by 2 qualified physicians.

    * The attending vascular surgeon will provide the primary assessment.
    * The confirmatory opinion must come from a fully licensed physician. (not a resident)
    * If anatomical considerations are invoked, the second physician may be a vascular surgeon, interventional radiologist, cardiologist, or vascular medicine specialist.
    * If medical co-morbidity is deemed the high risk aspect, then the confirmatory opinion may be obtained from an internist, family physician, cardiologist, vascular medicine, nephrologists, or vascular surgeon.
* Age >18 years and ability to understand the planned treatment
* Subject has read and signed the IRB approved Informed Consent form
* Patients for whom the following medication(s) is prescribed must have a one month stable baseline of appropriate/maximally tolerated therapy prior to enrollment: Plavix/asprin therapy, anticoagulation therapy, cholesterol lowering agent, and or blood pressure medication
* Hematocrit ≥ 28.0%, White Blood Cell count ≤ 14,000, Platelet count ≥ 50,000, Creatinine ≤ 2.0 mg / dL, INR ≤ 1.6 unless on Coumadin, or PTT <1.5 x control (to avoid bleeding complications) Patients on Coumadin will be corrected prior to the procedure and must have an INR<1.6 at the time of randomization/surgery.

Exclusion Criteria:

* Life expectancy <6 months due to concomitant illnesses
* History of bone marrow diseases (especially NHL, MDS) that prohibit transplantation
* Terminal renal failure with existing dependence on dialysis
* Known active malignancy or results outside of normal limits from the following tests: PAP, Chest X-ray, PSA, Mammogram, Hemoccult unless follow-up studies reveal patient to be cancer free..
* Poorly controlled diabetes mellitus (HgbA1C>10%)
* Medical risk that precludes anesthesia (conscious sedation), or ASA Class 5
* Life-threatening complications of the ischemia necessitating immediate amputation
* Uncorrected iliac artery occlusion on index side
* No Doppler signal in the foot (ABI =0)
* Extensive necrosis of the index limb or other conditions that make amputation inevitable (Rutherford Category 6)
* Active clinical infection being treated by antibiotics within one week of enrollment
* Treatment with immunosuppressant drugs (including Prednisone > 5 mg per day).
* Female who is pregnant or nursing, or of child bearing potential and is not using a reliable birth control method.
* Underwent a major open cardiovascular surgical procedure (carotid endarterectomy, arterial aneurysm or bypass surgery, or coronary artery bypass surgery) or a myocardial infarction within the 3 months prior to randomization
* Cerebrovascular accident within 6 months prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2007-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
To be determined by data from this feasibility study | 3 mos & 5 years

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of South Florida Department of Vascular Surgery at Tampa General, Tampa, Florida
  - Tufts Medical Center, Boston, Massachusetts
  - The Vascular Group at Albany Medical Center, Albany, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Roper St. Francis Hospital, Charleston, South Carolina
  - Methodist Hospital, Houston, Texas